CLINICAL TRIAL: NCT04111315
Title: Efficacy of Metamizole Versus Ibuprofen and a Short Educational Intervention Versus Standard Care in Acute and Subacute Low Back Pain: A Randomized, Factorial Trial
Brief Title: Efficacy of Metamizole Versus Ibuprofen and a Short Educational Intervention Versus Standard Care in Acute Low Back Pain
Acronym: EMISI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-01986
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: Pain medications; Non-opioid pain medications; Educational intervention
MeSH Terms: conditions — Low Back Pain | interventions — Dipyrone; Ibuprofen; Patient Education as Topic; Educational Status

STUDY DESIGN:
Intervention Model Description: Patients are assigned into one of the four groups metamizole + educational intervention metamizole + standard care ibuprofen + educational intervention ibuprofen + standard care Comparison (A): metamizole vs. ibuprofen for pain (NRS) at day 14 Comparison (B): short educational interventions vs. standard care for Disability (COMI) at day 42
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Comparison (A): participants, care provider, and Investigators will be blinded Comparison (B): Investigators will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- metamizole + educational intervention (Active Comparator): (A) Metamizole (Novalgin® Oblong tablets 0,5 g) orally three times daily 2 capsules for 4 days followed by an as needed regimen (days 4 - 42). The treatment duration will depend on the duration of pain. Patients are considered to be recovered when their pain is below 2 (NRS 0-10) on 2 consecutive days after they stopped the pain medication (end of treatment).
  (B) Educational short intervention: patients receive two leaflets with information non-specific LBP and exercises to alleviate LBP. Further, patients receive a 10-minute standardized telephone intervention during the first 4 treatment days.
  Interventions: Drug: Metamizole Sodium; Behavioral: Patient education
- metamizole + standard care (Active Comparator): (A) Metamizole (Novalgin® Oblong tablets 0,5 g) orally three times daily 2 capsules for 4 days followed by an as needed regimen (days 4 - 42). The treatment duration will depend on the duration of pain. Patients are considered to be recovered when their pain is below 2 (NRS 0-10) on 2 consecutive days after they stopped the pain medication (end of treatment).
  (B) Standard care will be prescribed by the GP.
  Interventions: Drug: Metamizole Sodium
- ibuprofen + educational intervention (Active Comparator): (A) Ibuprofen (Ibufen-L® tablets 500 mg) orally three times daily 2 capsules for 4 days followed by an as needed regimen (days 4 - 42). The treatment duration will depend on the duration of pain. Patients are considered to be recovered when their pain is below 2 (NRS 0-10) on 2 consecutive days after they stopped the pain medication (end of treatment).
  (B) Educational short intervention: patients receive two leaflets with information non-specific LBP and exercises to alleviate LBP. Further, patients receive a 10-minute standardized telephone intervention during the first 4 treatment days.
  Interventions: Drug: Ibuprofen 600 mg; Behavioral: Patient education
- ibuprofen + standard care (Active Comparator): (A) Ibuprofen (Ibufen-L® tablets 500 mg) orally three times daily 2 capsules for 4 days followed by an as needed regimen (days 4 - 42). The treatment duration will depend on the duration of pain. Patients are considered to be recovered when their pain is below 2 (NRS 0-10) on 2 consecutive days after they stopped the pain medication (end of treatment).
  (B) Standard care will be prescribed by the GP.
  Interventions: Drug: Ibuprofen 600 mg

INTERVENTIONS:
Drug: Metamizole Sodium — Novalgin® Oblong tablets 0,5 g 2-2-2
  Other Names: Metamizole
  Arms: metamizole + educational intervention; metamizole + standard care
Drug: Ibuprofen 600 mg — Ibufen-L® tablets 500 mg 2-2-2
  Other Names: Ibuprofen
  Arms: ibuprofen + educational intervention; ibuprofen + standard care
Behavioral: Patient education — Leaflet and phone call
  Other Names: Education
  Arms: ibuprofen + educational intervention; metamizole + educational intervention

SUMMARY:
The EMISI trial is a randomized, double blind, controlled trial (RCT) using a factorial design in patients with a new low back pain episode. The study aims to assess (A) whether metamizole, a non-opioid drug approved in Switzerland for pain treatment, is non-inferior to ibuprofen in a new episode of acute or subacute LBP and (B) whether a short educational intervention including evidence-based patient information is superior to usual care alone. Despite its increased use, the role of metamizole for the treatment of LBP is unclear and has so far not been systematically studied.

DETAILED DESCRIPTION:
Purpose Low back pain (LBP) is among the top three most common diseases worldwide resulting in a life with pain-related disability. In patients with persistent LBP over 3 months, the risk for chronic pain increases dramatically and effective interventions should aim to prevent pain persistence without overtreatment. Therefore, during an acute LBP episode, the most common recommendations are to use pain medication to alleviate pain and to keep patients physically active. Non-opioid and opioid pain medication is increasingly used to control pain. Despite the frequency of LBP, only few high-quality studies assessed the efficacy of pain medication. Since the 1990s, the use of opioid pain medication for non-cancer pain has soared and resulted in an epidemic of opioid dependence and abuse in the U.S. This, despite the fact that randomized clinical trials found little or no additional efficacy of opioids compared to non-opioid medication in LBP. Moreover, opioids are associated with potentially severe side-effects, including confusion, sedation, respiratory depression and dependence. Therefore, non-opioid pain medications that are safe and effective are urgently needed to control pain.

Non-steroidal anti-inflammatory drugs (NSAIDs) are considered to be effective for LBP and recommended by guidelines. However, adverse events including kidney injury and gastrointestinal bleeding, limit the use of NSAIDs in many patients. Metamizole is an effective non-opioid analgesic and antipyretic with a favorable gastrointestinal and renal safety profile and therefore, a valuable treatment option in many LBP patients with contraindications for NSAIDs. Metamizole has been increasingly used in many countries such as Germany, France, Spain, and Switzerland. Despite its increased use, the role of metamizole for the treatment of LBP is unclear and has so far not been systematically studied. This surprising lack of efficacy data may be due to an ongoing controversy over the risk of metamizole-associated agranulocytosis, a serious hematological adverse event. Even though the overall risk of agranulocytosis is increased compared to other drugs, it only occurs in a small proportion of susceptible patients and the overall safety profile of metamizole is still favorable compared to other analgesics such as NSAIDs or opioids, which carry their own specific risks.

Many patients have reservations against regular intake of pain medication and limit physical activity to keep pain manageable without medication, which is against the guidelines' recommendation. However, education to encourage activity may help to improve pain control and function as well. In a busy primary care practice extended educational sessions that have been shown to be effective are not feasible. A short educational intervention that provides evidence-based information on the nature of LBP and promotes physical activity may also improve outcome.

Objectives This study aims to assess (A) whether metamizole is non-inferior to ibuprofen in a new episode of acute or subacute LBP and (B) whether a short educational intervention including evidence-based patient information is superior to usual care alone.

Methods The EMISI trial is a randomized, double-blind, controlled trial (RCT) using a factorial design recruiting patients consulting general practitioners (GP) practices and the outpatient Division of the Department of General Internal Medicine at the University Hospital Bern, Switzerland. Patients are randomized into one of four groups (1:1:1:1): metamizole + educational intervention vs. metamizole + standard care vs. ibuprofen + educational intervention vs. ibuprofen + standard care. Patients assigned to the educational information will receive an information leaflet and a phone call by a member of the research team to discuss evidence based information on LBP. All patients will receive usual care provided by their GPs that includes additional pain medications and non-pharmacological measures at the GPs discretion.

The primary outcome (A) Comparison of ibuprofen vs. metamizole: change from baseline pain on the numeric rating scale (NRS) to day 14 (non-inferiority).

B) Comparison of the short intervention vs. usual care: change from baseline Core Outcome Measures Index (COMI) sum-score to 42 days follow-up (superiority).

Statistical analysis Analysis will include an intention-to-treat (ITT) and a per-protocol (PP) analysis for the comparison of the primary between metamizole and ibuprofen outcome (NRS change from baseline to follow-up at 14 days). Both analyses need to meet non-inferiority in order to claim success. The comparison of the primary outcome between the intervention and the usual care group (COMI change from baseline to day 42) will be performed according to intention-to-treat principle. Based on the sample size calculation for both interventions, 120 patients will be included into the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age 18 years or older
* Seeking care for new onset of non-specific or specific LBP (pain duration of less than 12 weeks LBP prior to the baseline visit)
* The GP plans to prescribe a non-opioid pain medication for pain control

Exclusion Criteria:

* Presence of red flags (serious neurological deficit requiring surgery, infection, vertebral fracture)
* Active malignancy and / or history of a (previous) hematologic disorder (anemia (hemoglobin < 10.0 g/L), neutropenia or agranulocytosis, thrombocytopenia),
* Known contraindications against the study medications: heart failure (NYHA III-IV), liver failure (liver cirrhosis, ascites), renal insufficiency (estimated glomerular filtration rate (eGFR) < 60 ml/min/1,73 m2) or previous acute kidney injury (AKI stage 2 according to the KDIGO definition), previous gastrointestinal ulcer, inflammatory bowel disease.
* Immune deficiency or under immunosuppressant treatment
* Current use of opioids
* Known intolerance to the study medication (i.e. previous acute allergic reaction to the study medication)
* Patients unable or unwilling to follow instructions or do not speak and are unable to read / understand German
* Patients unable to provide informed consent themselves
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow study procedures, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another study within the 30 days preceding the randomization and during the present study or previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Pregnancy: In women in the child bearing age a negative pregnancy test (urine or blood test as available in the primary care practice) before inclusion is required. Women who are not willing to use safe contraception (condom or birth control pill) during the course of the trial, intention to become pregnant during the trial, pregnancy, or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain improvement | Baseline to 14 days follow-up
  Change in pain on the numeric rating scale (NRS, range 0 (no pain) -10 (worst possible pain) points)
Disability | Baseline to 42 days follow-up
  Change in the Core Outcome Measures Index (COMI) sum-score (range 0-10). COMI sum score (0-10 points) is calculated by averaging the five domain scores (each on a 0-10 scale) for pain, back-related function, symptom-specific well-being, general quality of life and disability. Higher values represent a better or worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Maria M. Wertli, MD PhD, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Depending on the data privacy regulation, we aim to make individual participant data available opon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol will be made available upon request and will be shared as soon as the trial results are published.
Access Criteria: Contact the principal investigator

REFERENCES:
- [Background] Wertli MM, Flury JS, Streit S, Limacher A, Schuler V, Ferrante AN, Rimensberger C, Haschke M. Efficacy of metamizole versus ibuprofen and a short educational intervention versus standard care in acute and subacute low back pain: a study protocol of a randomised, multicentre, factorial trial (EMISI trial). BMJ Open. 2021 Oct 13;11(10):e048531. doi: 10.1136/bmjopen-2020-048531. PMID 34645660
- [Background] Jermini-Gianinazzi I, Blum M, Trachsel M, Trippolini MA, Tochtermann N, Rimensberger C, Liechti FD, Wertli MM. Management of acute non-specific low back pain in the emergency department: do emergency physicians follow the guidelines? Results of a cross-sectional survey. BMJ Open. 2023 Aug 4;13(8):e071893. doi: 10.1136/bmjopen-2023-071893. PMID 37541755